CLINICAL TRIAL: NCT02398201
Title: A Feasibility Study of Bezafibrate in Mitochondrial Myopathy
Brief Title: A Study of Bezafibrate in Mitochondrial Myopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7406
Record Dates: First submitted 2015-03-09; First posted 2015-03-25 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Bezafibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): Bezafibrate tablets (200-600mg) three times daily for 12 weeks.
  Interventions: Drug: Bezafibrate

INTERVENTIONS:
Drug: Bezafibrate — Bezafibrate 200mg-600mg three times daily for 12 weeks.
  Other Names: Bezalip

SUMMARY:
The purpose of this study is to gather preliminary data on whether bezafibrate can improve cellular energy production in mitochondrial disease.

Mitochondrial diseases are rare inherited disorders that arise due to deficient energy production within the cells of the body. Consequently, the typical clinical features arise in organs with high energy requirements. Mitochondrial disorders exhibit highly variable clinical effects, both between individuals and within families. Characteristic symptoms include muscle weakness (myopathy), hearing loss, migraine, epilepsy and stroke like episodes in addition to diabetes and heart problems. Mitochondrial disorders can therefore impact considerably on both quality of life and life expectancy. Despite this, no proven disease modifying treatments are available.

Pre-clinical studies have identified that several existing medications improve mitochondrial function. Of these, bezafibrate has the best supportive data and, because it is already licensed as a treatment for high blood fats, has a well characterised side effect profile.

The investigators will therefore conduct a feasibility study of bezafibrate in people with mitochondrial myopathy. Ten affected participants will be recruited and will receive a titrating course of bezafibrate three times daily for 12 weeks.

DETAILED DESCRIPTION:
Mitochondrial disorders are genetically determined metabolic diseases affecting approximately 1 in 5000 people. Current strategies for treating mitochondrial disorders are limited, and restricted to alleviating symptoms. A recently published Cochrane review did not identify any disease modifying treatments of proven benefit. There is therefore an urgent and currently unmet need for treatments that modify the underlying biochemical deficit and disease trajectory.

Improving deficient oxidative phosphorylation (OXPHOS) pathways through induction of mitochondrial biogenesis is a potential approach to the treatment of mitochondrial disorders. This involves stimulating transcription factors for both nuclear and mitochondrial genomes simultaneously in order to up-regulate respiratory chain (RC) gene expression. This role is fulfilled by peroxisome proliferator activated receptor (PPAR)-γ coactivator-1α (PGC-1α); a pivotal transcriptional co-factor widely considered the master regulator of mitochondrial biogenesis.

PGC-1α interacts with a number of transcription factors. These include α, β/δ and γ isoforms of the peroxisomal proliferator activated receptors (PPARs). This group of ubiquitously expressed nuclear receptors is activated by binding of fatty acids. Subsequently, transcription of genes involved in mitochondrial fatty acid oxidation is induced, thereby enabling cellular metabolic shift from glycolysis. Additionally, PGC-1α co-activates estrogen related receptor alpha (ERRα); nuclear respiratory factors (NRF) 1 and 2 (transcription factors bound to promoter regions of target nuclear genes involved in the respiratory chain); and TFAM (transcription factor A mitochondrial), which modulates mitochondrial DNA transcription and replication.

PGC-1α expression is induced through cold exposure, starvation and exercise. The PPARs, AMP-protein activated kinase (AMPK) and sirtuin 1 (Sirt1) also increase PGC-1α activity and provide a means through which this pathway can be pharmacologically manipulated. Indeed, several compounds have been identified that exert their effect in this way including: bezafibrate and the glitazones (PPAR agonists); metformin and AICAR (AMPK); and resveratrol (Sirt1). Of these, bezafibrate, glitazones and metformin have established relevance in diabetes and hyperlipidaemia. Their mechanism of action also provides a rationale for their use in other metabolic disorders such as obesity and mitochondrial disease.

Indeed,bezafibrate has shown promise as a disease modifying pharmaceutical agent in pre-clinical studies using both cellular and animal models of mitochondrial myopathy.

Cellular models of mitochondrial disease have demonstrated improvements in a variety of measures of mitochondrial function when grown in a bezafibrate enriched medium. This has included a cell line comparable to the specific patient group we propose to review in this feasibility study. Furthermore, a mouse model of mitochondrial myopathy has demonstrated improvement in clinically relevant outcomes including time to disease manifestation and life span.

This phase II, open label, non-randomised feasibility study aims to build on the work obtained in pre-clinical studies and provide proof of principle data in humans affected with the most common form of mitochondrial muscle disease. This study is not designed to provide proof of efficacy. However, should bezafibrate exert a demonstrable molecular effect here, the investigators anticipate the need for larger, randomised trials of bezafibrate in the future. An additional aim of this feasibility study, is therefore obtaining the relevant data to determine how many patients the investigators would need in a larger trial; and what biochemical and clinical measurements the investigators would use to determine drug effect in such a trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* The participant is willing and able to given informed consent for participation
* Confirmed mt.3243A>G mutation
* Evidence of myopathy
* Stable dose of current regular medication for at least 4 weeks prior to trial entry
* Not already taking fibrates
* No evidence of liver impairment
* Normal renal function with a creatine clearance of >60ml/minute
* In the investigator's opinion is willing and able to comply with all trial requirements
* Willingness to allow General Practitioner and Hospital Consultant to be notified of participation in the trial

EXCLUSION CRITERIA:

* contraindication to MRI scanning
* Unstable or poorly controlled diabetes, as determined by the investigator. Participants assigned to group 2 dosing with diabetes (insulin or non-insulin dependent) or glucose intolerance who are unwilling or unable to monitor blood glucose levels during the 12 week treatment period
* Previous episode of rhabdomyolysis
* History of sensitivity to fibrates
* History of gallbladder disease (with or without cholelithiasis)
* Liver impairment or disease
* Alcohol misuse
* Nephrotic syndrome
* Untreated hypothyroidism
* Use of other medication interacting with bezafibrate
* A female participant who is pregnant, lactating or planning pregnancy during the course of the trial; or a male participant who is planning to conceive with their female partner.
* Elective or emergency surgery in the 12 weeks prior to screening visit
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial
* Any other significant disease or disorder which, in the opinion of the investigator, may put the participant at risk; may influence the result of the trial; or will compromise the individual's ability to participate in the trial.
* Participants who have taken part in another research trial involving an investigational medicinal product in the last 12 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Change in Respiratory Chain Enzyme Activity | baseline and 12 weeks

SECONDARY OUTCOMES:
Change in citrate synthase | baseline and 12 weeks
Change in mitochondrial DNA copy number | baseline and 12 weeks
Change in COX negative fibres | baseline and 12 weeks
Change in serum Fibroblast Growth Factor-21 concentration | baseline, 3, 6, 9, 12 weeks
Change in PGC-1alpha concentration | baseline, 3, 6, 9, 12 weeks
Change in micro-RNA expression pattern | baseline, 3, 6, 9, 12 weeks
Change in cardiac 31P-MRS | baseline and 12 weeks
  We will specifically analyse ATP production and muscle phosphocreatine pre and post bezafibrate
Change in cardiac cine MRI | baseline and 12 weeks
  We will analyse LV (left ventricular) torsion pre and post bezafibrate
Change in skeletal muscle 31P-MRS | baseline and 12 weeks
  We will analyse ATP production, muscle phosphocreatine, t1/2 PCR (phosphocreatine), muscle lipid content and volume.
Change in IPAQ (international physical activity questionnaire) score | baseline, 6 and 12 weeks
Change in accelerometry | baseline, 6 and 12 weeks
Change in Timed Up and Go (TUG) time | baseline, 6 and 12 weeks
Change in NMDAS (Newcastle Mitochondrial Disease Adult Scale) score | baseline, 6 and 12 weeks
Change in heteroplasmy level | baseline and 12 weeks
  measured in blood, urine and muscle
Change in NMQ (Newcastle Mitochondrial Disease Quality of Life) Score | baseline, 6 and 12 weeks
Change in Fatigue Impact Scale score | baseline, 6 and 12 weeks
Number of Adverse Events | 0,1,2,3,4,5,6,7,8,9,10,11,12,13,14 weeks
  Adverse events will be captured every week with opportunistic capture between visits as required.
Change in Full Blood Count | 0,1,2,3,4,5,6,7,8,9,10,11,12 weeks
  White cell count; Haemoglobin; Platelet count
Change in Urea & Electrolytes | 0,1,2,3,4,5,6,7,8,9,10,11,12 weeks
  Sodium; Potassium; Urea; Creatinine;
Change in Liver Function Tests | 0,1,2,3,4,5,6,7,8,9,10,11,12 weeks
  Alkaline Phosphatase, Alanine Transferase, Aspartate Aminotransferase, Gamma Glutamyl Transferase
Change in Creatine Kinase | 0,1,2,3,4,5,6,7,8,9,10,11,12 weeks
Change in Prothrombin Time | 0,1,2,3,4,5,6,7,8,9,10,11,12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Chinnery, MBBS, PhD, Principal Investigator — Newcastle Univeristy
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided